CLINICAL TRIAL: NCT01875016
Title: Endocardial Catheter CRyo-Ablation of Septal Hypertrophy for Hypertrophic Obstructive Cardiomyopathy
Brief Title: CRyo-Ablation to Treat Patients With HOCM.
Acronym: CRASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, MEDINA AHARON, Head of EP Unit, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRASH
Record Dates: First submitted 2013-06-04; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: HOCM, Hypertrophic Obstructive Cardiomyopathy
Keywords: Cryo ablation; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: CRyo-Ablation to Treat HOCM. — CRyo-Ablation to Treat Patients With HOCM.

SUMMARY:
The purpose of the study is to perform endocardial catheter CRyo-Ablation to relieve the LVOT obstruction in patients with Hypertrophic Obstructive Cardiomyopathy.

The investigators hypothesize that the investigators will be able to reduce > 50% of the initial LVOT gradient. This will be considered as a successful procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 years of age
2. The patient has left ventricular outflow tract obstruction with hypertrophic obstructive cardiomyopathy
3. The patient is on optimal medication
4. The patient is not eligible for/failed/refused alcohol ablation
5. The patient is not eligible for/failed/refused myectomy
6. The patient is willing to participate in the study and has signed informed consent
7. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved be the appropriate medical ethics committee.

Exclusion Criteria:

1. Pregnant or nursing patients Female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test
2. Patient has history of or known impaired renal function (Serum creatinine >2.0 mg/dL or 177 µmol/l) or on dialysis
3. Patient has a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated
4. Patient has a known hypersensivity or contraindication to aspirin, both heparin and bivalirudin, clopidogrel and/or contrast sensitivity/allergy that cannot be adequately pre-medicated
5. Patient has other medical illness not related to the hypertrophic cardiomyopathy (e.g., cancer, known malignancy, or cognitive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with limited life expectancy (i.e., less than 1 year)
6. Subject is enrolled or intended to participate in any concurrent drug and/or device study, which would confound the results of this trial as determined by the investigator, during the course of this clinical study
7. Subjects meets the exclusion criteria required by local low (e.g. age, pregnancy, breast-feeding, etc)
8. Subject is anticipated not being able to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Acute and long term reduction of initial LVOT gradient | Post procedure and up to 12 months follow up

SECONDARY OUTCOMES:
Number of patients with procedure related complications. | During the procedure untill discharge.

REFERENCES:
- [Background] Keane D, Hynes B, King G, Shiels P, Brown A. Feasibility study of percutaneous transvalvular endomyocardial cryoablation for the treatment of hypertrophic obstructive cardiomyopathy. J Invasive Cardiol. 2007 Jun;19(6):247-51. PMID 17541123
- [Background] Lawrenz T, Borchert B, Leuner C, Bartelsmeier M, Reinhardt J, Strunk-Mueller C, Meyer Zu Vilsendorf D, Schloesser M, Beer G, Lieder F, Stellbrink C, Kuhn H. Endocardial radiofrequency ablation for hypertrophic obstructive cardiomyopathy: acute results and 6 months' follow-up in 19 patients. J Am Coll Cardiol. 2011 Feb 1;57(5):572-6. doi: 10.1016/j.jacc.2010.07.055. PMID 21272748